CLINICAL TRIAL: NCT04505813
Title: A Phase 1 / 2 Study to Evaluate the Safety and Tolerability of Adoptively Transferred Autologous T Cells in Patients With Relapsed Refractory Multiple Myeloma
Brief Title: Antigen-specific T Cell Therapy for Patients With Relapsed Refractory Multiple Myeloma
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: NexImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEXI-002-01
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Relapsed Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Evaluation Phase (Experimental): Treatment with NEXI-002 T cells, derived from PBMCs of the patient
  Interventions: Biological: NEXI-002 T Cells
- Dose Expansion Phase (Experimental): Dose Expansion Phase to further define the safety, tolerability and initial anti-tumor efficacy of the NEXI- 002 T cell product at the dose established from the Safety Evaluation Phase.
  Interventions: Biological: NEXI-002 T Cells

INTERVENTIONS:
Biological: NEXI-002 T Cells — The NEXI-001 T cell product will be administered as a single IV infusion to patients within 72 hours after completing LD therapy.

SUMMARY:
This Research study is being done to characterize the safety, tolerability, and preliminary antitumor activity of the NEXI-002 T cell product (a new experimental therapy), which contains populations of CD8+ T cells targeting multiple Myeloma associated antigen peptides in patients with relapsed refractory multiple myeloma (MM).

The study will enroll patients with MM who have relapsed or are refractory to standard lines of treatment.

The enrolled patients will undergo bridging therapy for the purposes of disease control while the NEXI-002 T cell product is being manufactured. Choice of bridging therapy administered will be per the Investigator's discretion, but is limited to acceptable agents as specified in the protocol. Bridging therapy will be administered prior to lymphodepleting (LD) therapy, with the last dose of the bridging therapy administered ≥ 14 days prior to initiation of LD therapy. Within 72 hours after completing LD therapy, patients will receive a single IV infusion of the NEXI-002 T cell product.

DETAILED DESCRIPTION:
The NEXI-002 is an adoptive cellular therapy product which contains populations of antigen-specific CD8+ T cells. The antigen-specific CD8+ T cells in the NEXI-002 T cell product are derived from Peripheral Blood Mononuclear Cells (PBMC) obtained from the patient. During the manufacturing process, these cells are primed and expanded ex vivo using nano-size artificial Antigen Presenting Cells (aAPC) loaded with five leukemia associated antigen peptides in combination with a proprietary T cell enrichment and expansion process.

The NEXI-002 T cell product is restricted to patients that are HLA-A2.01 allele positive for this study.

There are two parts to this study, a Safety Evaluation Phase and a Dose Expansion Phase. The Safety Evaluation Phase will determine the safety and tolerability of a single dose of NEXI-002 T cell product, and will consist of Dose Escalation at two dose levels - each with cohorts of three patients.

When all three patients at Dose Level 1 have dosed and cleared the DLT period, three additional patients will be enrolled at Dose Level 2. When three patients have cleared the DLT period at the highest dose level, that dose will be advanced to the Dose Expansion Phase. The Dose Expansion Phase will enroll up to 16 additional patients to further define the safety and evaluate the initial anti-tumor efficacy of the NEXI- 002 T cell product at the dose established from the Safety Evaluation Phase.

All patients will enter a Post-Treatment Follow-Up period after infusion of the NEXI- 002 T cell product. During this phase, all patients will be monitored for AEs and followed for anti-leukemia response until the end of study visit is complete (up to one year).

Additional assessments for safety, disease status, and other secondary and exploratory endpoints will also be monitored during the follow-up period.

All patients will be followed for overall survival (OS) from time of disease progression until the last visit of the last patient. During this time, patients will be followed via telephone or other electronic contact at 12 week intervals for monitoring of OS.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent and documentation of informed consent prior to initiation of any study-related tests or procedures that are not part of standard-of-care for the patient's disease. Patients must also be willing and able to comply with study procedures, including the acquisition of specified research specimens
2. Age ≥ 18 years old & life expectancy > 3 months
3. Expression of HLA-A*0201 as determined by high resolution sequence-based typing method
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with exception of ECOG > 1 if related to recent bone fracture
5. Patients must have confirmed diagnosis of MM
6. Have identified relapsed/refractory disease which includes:

   1. Previous therapy consisting of at least three (3) standard regimens, including a proteasome inhibitor, IMiD, or anti-CD38 targeting therapy.

      Note: Induction therapy, autologous stem cell transplantation (ASCT) & maintenance therapy if given sequentially without intervening progressive disease (PD) are considered one 'regimen'
   2. Refractory MM may be defined as disease that is refractory to treatment while on therapy or that shows progression within 60 days of the last therapy.
7. Have measurable disease as defined by:

   1. Serum M protein ≥ 0.5 g/dL
   2. Urine M protein ≥ 200 mg/24hr
   3. Serum free light chains (FLC) ≥ 10 mg/dL with abnormal FLC ratio Note: Patients with IgA MM in whom serum protein electrophoresis (sPEP) is deemed unreliable, due to co-migration of normal serum proteins with the paraprotein in the β region, may be considered eligible as long as total serum IgA level is > normal range.
8. Acceptable laboratory parameters as follows:

   1. AST/ALT ≤ 2.5 × ULN
   2. Total bilirubin ≤ 1.5 × ULN, except patients with Gilbert's syndrome, who may enroll if the conjugated bilirubin is within normal limits
   3. Serum creatinine ≤ 2.5 mg/dL or estimated creatinine clearance (CL) ≥ 30 mL/min & not dialysis-dependent
   4. ALC > 1000 cells/µL
9. Recovery to Grade 1 or baseline of non-hematologic toxicities from prior treatments, excluding alopecia & Grade 2 peripheral neuropathy
10. Female patients of childbearing potential must test negative for pregnancy at enrollment and during the study. Sexually active women of child-bearing potential, unless surgically sterile, must be willing to use a highly effective method of birth control defined as those which result in a low failure rate (i.e., less than 1% per year) such as implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs) or vasectomized partner
11. Male patients with partners of childbearing potential must be either vasectomized or agree to use a condom in addition to having their partners use another method of contraception resulting in a highly effective method of birth control defined as those which result in a low failure rate (i.e., less than 1% per year) such as implants, injectables, combined oral contraceptives, or IUDs. Patients should not have sexual intercourse with females who are either pregnant or lactating without double-barrier contraception • Is not pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the prescreening or screening visit through one year from administration of NEXI-002 T cells

Exclusion Criteria:

1. Have active cerebral or meningeal disease related to the underlying malignancy
2. Have hemolytic anemia, plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome, amyloidosis, plasmacytoma, significant autoimmune or other malignant disease
3. History of allogeneic hematopoietic stem cell transplantation
4. Have active or uncontrolled infections with positive cultures and/or requiring treatment with IV anti-infective agents
5. Echocardiogram or MUGA with left ventricular ejection fraction < 45%
6. History of clinically significant cardiovascular disease including but not limited to:

   1. Myocardial infarction or unstable angina within the 6 months prior to the initiation of study
   2. Stroke or transient ischemic attack within 6 months prior to initiation of study
   3. Clinically significant cardiac arrhythmia
   4. Uncontrolled hypertension: systolic blood pressure (SBP) > 180 mmHg, diastolic blood pressure (DBP) > 100 mmHg
   5. Congestive heart failure (New York Heart Association [NYHA] class III-IV)
   6. Pericarditis or clinically significant pericardial effusion
   7. Myocarditis
7. Clinically significant pulmonary compromise, including a requirement for supplemental oxygen use to maintain adequate oxygenation
8. Eligible patients will not be on any steroids ≥10 mg per day prednisone or equivalent or other immunosuppressants such as tacrolimus, cyclosporine, etc.

   a. Intermittent topical, inhaled or intranasal corticosteroids are allowed
9. History of symptomatic deep vein thrombosis (DVT) or pulmonary embolism (PE) requiring systemic anticoagulation within 6 months before enrollment
10. History of autoimmune disease (e.g., Crohn's, rheumatoid arthritis, systemic lupus erythematosus, etc.) resulting in end organ injury or requiring systemic immunosuppression / systemic disease modifying agents within the last 2 year prior to enrollment. Subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and subjects with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for the study
11. Human immunodeficiency virus (HIV) seropositive; HIV testing within 2 years of enrollment
12. Seropositive for and with evidence of active viral infection with hepatitis B virus (HBV). Patients who are hepatitis B surface antigen (HBsAg) negative and HBV viral DNA negative are eligible

    1. Patients who had HBV but have received an antiviral treatment and show non-detectable viral DNA for 6 months are eligible
    2. Patients who are seropositive because of HBV vaccine are eligible
13. Seropositive for and with active viral infection with hepatitis C virus (HCV)

    a. Patients who had HCV but have received an antiviral treatment and show no detectable HCV viral DNA for 6 months are eligible
14. Second primary invasive malignancy that has not been in remission for more than 2 years. Exceptions that do not require a 2-year remission include: non-melanoma skin cancer; carcinoma in situ (cervix, bladder, breast, etc.) or squamous intraepithelial lesion on Pap smear; localized prostate cancer (Gleason score < 6); or resected melanoma in situ
15. History of trauma or major surgery within 4 weeks prior to the initiation of study
16. Any serious underlying medical or psychiatric condition that would impair the ability of the patient to receive or tolerate the planned treatment and follow up
17. Known hypersensitivity to any component of NEXI-002 T cells, cyclophosphamide, fludarabine or tocilizumab
18. Vaccination with any live virus vaccine within 6 weeks prior to the initiation of study treatment. Inactivated annual influenza vaccination is allowed
19. Dementia or altered mental status that would preclude understanding and rendering of informed consent
20. History of seizures, aphasia, psychosis or other chronic clinically significant neurologic disorders

    a. Patients with remote history of seizures that are well controlled on anti-seizure medications and without any seizure episode for 6 months are eligible
21. Any issue that in the opinion of the investigator, would contraindicate the patient's participation in the study or confound the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events of Special Interest (AESIs) events | 1 year
  1) Dose Limiting Toxicities (DLTs).
Progressive Free Survival | At 12 months
  Median Progressive free Survival (PFS)
Overall Response Survival (Rate) | At 12 months
  Overall Response Rate (ORR)
Survival | At 12 months
  Overall Survival (OS)
Adverse events (AEs) Reporting | At year 1
  Incidence of TEAEs leading to study withdrawal
Adverse Events of Special Interest (AESIs) events (AEs) Reporting | at year 1
  Cytokine Release Syndrome (CRS)
Adverse Events of Special Interest (AESIs)events (AEs) Reporting (ICANS) | at year 1
  Immune effector Cell-Associated Neurotoxicity Syndrome (ICANS)
Adverse Events of Special Interest (AESIs)events (AEs) Reporting-TEAEs | At year 1
  For Incidence of TEAEs and serious TEAEs (Treatment-emergent adverse events (TEAEs) are defined as those AEs that started on or after LD therapy or that worsened after LD therapy.
Adverse Events of Special Interest (AESIs)events (AEs) Reporting-Infusion Reactions | At year 1
  Infusion Related Reactions (IRR)

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Jones, Study Chair — NexImmune
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Advent Health Medical Group Blood & Marrow Transplant, Orlando, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No